CLINICAL TRIAL: NCT06075368
Title: A Prospective, Multicenter, Observational Study to Evaluate the Efficacy and Safety of GENOSS SES in Patients With Acute Coronary Syndrome
Brief Title: Efficacy and Safety of GENOSS® SES in Patients With Acute Coronary Syndrome (GENOSS ACS)
Acronym: GENOSS ACS
Status: Active, not recruiting | Type: Observational
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-DS0501-10
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-02

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention
Keywords: ACS
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GENOSS® DES Sirolimus Eluting Coronary Stent System / B03300.20, class [4]: Patients with acute coronary syndrome treated with the GENOSS SES
  Interventions: Device: GENOSS Sirolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: GENOSS Sirolimus Eluting Coronary Stent System — The GENOSS SES is a novel, biodegradable, polymer-coated, sirolimus-eluting stent with a cobalt chromium stent platform and thin strut.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of the GENOSS SES in patients with acute coronary syndrome (ACS) in real-world pratice.

DETAILED DESCRIPTION:
The Genoss SES is a novel, biodegradable, polymer-coated, sirolimus eluting stent with a cobalt-chromium stent platform and thin strut. Although the efficacy and safety of this stent have been previously investigated, real-world clinical outcomes data are lacking. Therefore, the objective of this prospective, multicenter study was to evaluate the clinical efficacy and safety of the Genoss SES in acute coronary syndrome (ACS) patients undergoing percutaneous coronary intervention.

The Genoss SES study is a prospective, single-arm, observational study for evaluation of clinical outcomes after Genoss SES implantation in ACS patients undergoing percutaneous coronary intervention from 10 sites in South Korea. The primary endpoint was a device-oriented composite endpoint (DOCE), defined as a composite of cardiac death, target vessel-related myocardial infarction (MI), and clinically indicated target lesion revascularization (TLR) at 10 months.

ELIGIBILITY:
<Inclusion Criteria>

1. Patients of 19 and over
2. Patients with acute coronary syndrome treated with GENOSS SES
3. Participants who voluntarily decide to participate in this clinical trial, agree to the study protocol and clinical follow-up plan, and provide written informed consent as study participants.

<Exclusion Criteria>

1. Patients who are contraindicated in the use of heparin, aspirin, clopidogrel, sirolimus, cobalt chromium and contrast agents

   - However, patients with hypersensitivity to contrast agents may be eligible if it can be controlled by steroids and pheniramine. Patients with known anaphylaxis are excluded
2. Patients who are pregnant or planning to become pregnant
3. Patients scheduled to undergo surgery requiring the discontinuation of antiplatelet agents within 12 months from registration.
4. Patients with a life expectancy of less than 1 year
5. Patients who presented with cardiogenic shock at admission and are predicted to have a low chance of survival based on medical judgment.
6. Patients who have already received treatment with another DES (Drug Eluting Stent), BVS (Bioresorbable Vascular Scaffolds), or BMS (Bare Metal Stent) at the time of registration.
7. Patients currently participating in a randomized controlled trial involving medical devices.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome treated with the GENOSS SES
Sampling Method: Non-Probability Sample
Enrollment: 757 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Device-oriented composite endpoint | 12 months after the procedure
  DOCE is defined as a composite of cardiac death, target vessel-related myocardial infarction (TV-MI) and clinically indicated target-lesion revascularization (TLR).

SECONDARY OUTCOMES:
Target lesion failure (TLF) | 3 years after the procedure
  Target lesion failure (TLF) is defined as a composite of cardiac death, target vessel-related myocardial infarction (TV-MI) and clinically indicated target-lesion revascularization (TLR).
Target vessel failure (TVF) | 3 years after the procedure
  Target vessel failure (TVF) is defined as a composite of cardiac death, target vessel-related myocardial infarction (TV-MI) and clinically indicated target-vessel revascularization (TVR).
All-cause death | 3 years after the procedure
Cardiac death | 3 years after the procedure
All-cause death and any myocardial infarction | 3 years after the procedure
Cardiac death and target vessel-related myocardial infarction | 3 years after the procedure
Target vessel revascularization (TVR) | 3 years after the procedure
Target lesion revascularization (TLR) | 3 years after the procedure
Stent thrombosis | 3 years after the procedure

OTHER OUTCOMES:
Safety evaluation | 1 month, 12 months, 2 years, 3 years after the procedure
  Occurrence of stent-related events (cardiac death, myocardial infarction, stent thrombosis, bleeding, etc.) and any damage or complications that are believed to be related to the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No